CLINICAL TRIAL: NCT06646107
Title: Adherence to Mediterranean Diet in Type 1 Diabetes Initiating Minimed 780G: Glucose Metrics vs Insulin Metrics, is There a Difference
Status: Recruiting | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, VAIA LAMBADIARI, Professor of Internal Medicine-Endocrinology, Attikon Hospital
Other Study IDs: MED_TYPE 1
Record Dates: First submitted 2024-10-13; First posted 2024-10-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Type1diabetes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Type 1 Diabetes Mellitus: patients aged >12 years old with T1DM who are on multiple daily injections or insulin pump and are scheduled to start using MiniMed 780G
  Interventions: Device: MInimed 780G

INTERVENTIONS:
Device: MInimed 780G — Minimed 780G HCL system (Metronic, Northridge, Ca, USA) is ConformitèEuropëenne(CE)-marked and includes additional functionality aiming to provide further protections from high glucose levels. When the system is used in Auto Mode automatically calculate the insulin dose based on information received from CGM. Signals are converted by the transmitter to sensor glucose values. Sensor values are then transmitted to the insulin pump. Sensor glucose and insulin delivery data are stored by the pump and may be uploaded. The HCL system can be programmed to automatically calculate insulin doses (both basal insulin and correction boluses) based on information received from CGM780G and the adherence to MD.

SUMMARY:
In this observaltional study, 240 patients aged >12 years old with T1DM who are on multiple daily injections or insulin pump and are scheduled to start using MiniMed 780G system will be included.We aim to compare patients' adherence to Mediterranean diet (MD) before and 12 weeks after initiation of MiniMed 780G and its association with CGM and insulin metrics, as well as anthropometric measurements, BMI, body composition, lipid levels, blood pressure and gut microbioma. Moreover, at baseline, at six and 12 months, markers of endothelial and cardiovascular function will be also assessed and associated with the use of Minimed 780G and the adherence to MD.

DETAILED DESCRIPTION:
This observational study will include 240 participants (80 participants per country) from IGI region (Italy, Greece and Israel), children adolescents and young adults (12> years old) with T1D that are on multiple daily injections or insulin pump and are scheduled to start using MiniMed 780G system. After a 7-day run-in period, participants will be evaluated with food intake log and adherence to Meditteranean Diet (MD) with PREDIMED questionnaire. One hour session on MD and healthy impact on Diabetes will be provided to all participants and will be assigned to initiate MiniMed 780G and followed for 12 weeks. HbA1c, CGM and Insulin Metrics, anthropometric measurements, body composition, blood pressure and lipid leves as well a gut microbioma will be performed at baseline and 12 weeks, after MiniMed 780G initiation. A 7-day food diary logbook will be collected to identify the amount and type of the food at baseline and at the end of the study. At baseline, at 6 and at 12 months, markers of endothelial and cardiovascular function will also be assessed. An extension phase will include additional 3 and 6, which concludes one year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes >1 year prior to consent date. Diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not required.
2. HbA1c < 12.5%
3. Age >7years at the initiation of the system
4. Multiple Daily Injections (Basal Bolus therapy) with Total daily insulin use of great than 8.0 units per day over a 1-week period
5. Clinically able to start the AHCL system
6. History of 3 clinic visits in the last year

Exclusion Criteria:

1. Diabetic Ketoacidosis in the 6 months prior to screening visits

-

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children adolescents and young adults (12> years old) with T1D that are on multiple daily injections or insulin pump and are scheduled to start using MiniMed 780G system.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Hba1c | Baseline, 3 months
  Differences in HbA1c at baseline and 3 months after the initiation of MiniMed 780G
Changes in TIR | Baseline, 3 months
  Changes in TIR at baseline and 3 months after the initiation of MiniMed 780G
Changes in TBR | Baseline, 3 months
  Changes in TBR at baseline and 3 months after the initiation of MiniMed 780G
Changes in TAR | Baseline, 3 months
  Changes in TAR at baseline and 3 months after the initiaton of MiniMed 780G
Changes in bolus doses | Baseline, 3 months
  Changes in bolus dosed at baseline and 3 months after the initiation of MiniMed 780G
Changes in basal doses | Baseline, 3 months
  Changes in basal doses at baseline and 3 months after the initiation of MiniMed 780G
Changes in autocorrection doses | Baseline, 3 months
  Changes in autocorrection doses between baseline and 3 months after the initiation of MiniMed 780G:

SECONDARY OUTCOMES:
Changes in pulse wave velocity(m/s) | Baseline, 6 months, 12 months
  Changes in pulse wave velocity at baseline and at 6 and 12 months after the initiation of MiniMed 780G
Changes in endothelial glycocalyx thickness (μm) | Baseline, 6 months, 12 months
  Changes in endothelial glycocalyx thickness at baseline and at 6 and 12 months after the initiation of MiniMed 780G
Changes in global longidutinal strain (%) | Baseline, 6 months, 12 months
  Changes in global longidutinal strain at baseline and at 6 and 12 months after the initiation of MiniMed 780G
Changes in CAP (dB/m) | Baseline, 6 months, 12 months
  Changes in liver steatosis at baseline and at 6 and 12 months after the initiation of MiniMed 780G as assessed by the measurement of CAP. CAP score will be used as an index of liver fat content, with normal values being < 238 dB/m. <237 dB/m (S0, no steatosis), 237 -259 dB/m (S1, mild steatosis), 259 -291 dB/m (S2, moderate steatosis), and 291 -400 dB/m (S3,severe steatosis). E score will be used as an index of liver fibrosis. The cut-off values for fibrosis (F) were as follows:(1) <5.5 kPa (F0, no fibrosis), (2) 5.5-8.0 kPa (F1, mild fibrosis), (3) 8.0-10.0 kPa (F2, moderate fibrosis),(4) 11.0-16.0 kPa (F3, severe fibrosis), and (5) >16.0 kPa (F4, cirrhosis).
Changes in gut microbioma | Baseline,3 months
  Changes in gut microbioma at baseline and at 3 months after the initiation of MiniMed 780G.
Changes in coronary flow reserve | Baseline, 6 months, 12 months
  Changes in coronary flow reserve at baseline, at six months and at 12 months after the initiation of MiniMed 780G.
Changes in central aortic blood pressure (mmHg) | Baseline, 6 months, 12 months
  Changes in central aortic blood pressure at baseline and at 6 and 12 months after the initiation of MiniMed 780G.
Changes in Ε score (Kpa) | Baseline, 6 months, 12 months
  Changes in liver steatosis at baseline and at 6 and 12 months after the initiation of MiniMed 780G as assessed by E score. E score will be used as an index of liver fibrosis. The cut-off values for fibrosis (F) were as follows:(1) <5.5 kPa (F0, no fibrosis), (2) 5.5-8.0 kPa (F1, mild fibrosis), (3) 8.0-10.0 kPa (F2, moderate fibrosis),(4) 11.0-16.0 kPa (F3, severe fibrosis), and (5) >16.0 kPa (F4, cirrhosis).

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon University General Hospital, Chaïdári, Greece

IPD SHARING:
Plan to Share IPD: Undecided